CLINICAL TRIAL: NCT02559752
Title: Computer-based Neurocognitive Assessment in Children With Central Nervous System Tumors Receiving Proton Beam Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201509033
Record Dates: First submitted 2015-09-17; First posted 2015-09-24 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Central Nervous System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm 1: NIH Toolbox Cognitive Battery testing: * This study will use the NIH Toolbox Cognitive Battery computer testing software to investigate the cognitive outcomes in children with CNS tumors receiving PBRT.
  * Participants recruited for the study will complete one 45-minute testing session prior to the completion of the first week of radiation therapy.
  * They will then complete serial tests 6-12 months after the completion of PBRT and then yearly thereafter.
  Interventions: Other: NIH Toolbox Cognitive Battery

INTERVENTIONS:
Other: NIH Toolbox Cognitive Battery — * For ages 4 to 7 years, the NIH Toolbox Early Childhood Battery will be administered. This test includes the Picture Vocabulary, Flanker Inhibitory Control and Attention, Dimensional Change Card Sort, and Picture Sequence Memory measures to evaluate language, executive function, attention, and episodic memory, respectively.
  * For patients age 8 years or older, the administered battery will consist of the aforementioned tests in addition to Oral Reading Recognition, Pattern Comparison Processing Speed, and List Sort Working Memory tests. Results will include scores for each individual measure. In addition, each cognition battery provides composite scores, which allow for general interpretation/evaluation of overall cognitive functioning.

SUMMARY:
This study will explore neurocognitive performance in pediatric brain tumor patients receiving proton beam radiation therapy (PBRT). The investigators goal is to gather baseline neurocognitive testing prior to the completion of the first week of radiation therapy along with follow-up testing 6-12 months after the completion of radiation and serial annual testing thereafter. With these data the investigators plan to evaluate the effects of PBRT on neurocognitive performance as it relates to patients' age at diagnosis, tumor location, and radiation dose. Modeling studies have demonstrated that PBRT could improve neurocognitive outcomes, but there is a paucity of prospectively-collected patient data. The investigators are uniquely positioned to address this important question given the busy pediatric central nervous system (CNS) tumor service, the delivery of proton therapy at the S. Lee Kling Proton Therapy Center at Barnes-Jewish Hospital, and the multi-disciplinary research team with extensive experience into the late effects of therapy as it relates to neurocognition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary CNS tumor or diagnosis of metastatic disease to the CNS with an expected overall survival of > 1 year. Any prior treatment (chemo, XRT, or surgery) is allowed.
* Planning to receive PBRT to treat the CNS tumor. Patients who have already received PBRT for this disease may also be enrolled provided they completed the NIH Toolbox Cognitive Battery prior to the first week of radiation therapy.
* Between 4 and 21 years of age (inclusive).
* Life expectancy of at least one year.
* Absence of visual impairment that would impede computer testing.
* No secondary health conditions that would impact cognitive functioning (e.g. psychiatric or developmental disability unrelated to cancer).
* Able to understand and willing to sign IRB-approved written informed consent document (or signature of legally authorized representative).

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants seen at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-10-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of obtaining serial computer-based neurocognitive testing as measured by an acceptance rate of 60% of eligible patients. | At the completion of enrollment of all patients (estimated to be 9 years)
  The acceptance rate will be a proportion of those who consent to participation over the total number of eligible and approached participants. The 60% acceptance rate is chosen because previous behavioral science intervention study participation in pediatric hematology and oncology ranges from 42% to 90%.
Feasibility of obtaining serial computer-based neurocognitive testing as measured by an implementation rate of 80% among survivors | 12 months
  An implementation rate will be calculated by tracking the proportion of consented participants who complete at least two assessments in the first year of follow up. The primary length of time for implementation is in the first 12 months, but the rate of implementation will be tracked for up to five years for each participant. This is consistent with a two-staged assessment from Butler's remediation trial.
Feasibility of obtaining serial computer-based neurocognitive testing as measured by an implementation rate of 80% among survivors | 5 years
  An implementation rate will be calculated by tracking the proportion of consented participants who complete at least two assessments in the first year of follow up. The primary length of time for implementation is in the first 12 months, but the rate of implementation will be tracked for up to five years for each participant. This is consistent with a two-staged assessment from Butler's remediation trial.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Perkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu